CLINICAL TRIAL: NCT03313180
Title: An Open-label Extension Trial of the Long Term Safety of Nintedanib in Patients With 'Systemic Sclerosis Associated Interstitial Lung Disease' (SSc-ILD)
Brief Title: A Trial to Evaluate the Safety of Long Term Treatment With Nintedanib in Patients With Scleroderma Related Lung Fibrosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1199-0225; 2016-003403-66 (EudraCT Number)
Expanded Access: NCT03843892 (Approved for marketing)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nintedanib (Experimental): Patients with Systemic Sclerosis associated Interstitial Lung Disease (SSc-ILD) who took part in the parent trials 1199.214 (Nintedanib or Placebo) or 1199-0340 (Nintedanib). Patients continued in this trial and received Nintedanib 150 mg (milligram) twice daily (bid) unless they had reduced their dose to 100 mg bid trial medication (Nintedanib or Placebo) in the parent trial.
  Patients receiving 100 mg bid trial medication at the end of the parent trial could receive either Nintedanib 100 mg bid or 150 mg bid at the discretion of the investigator.
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Administered twice daily
  Other Names: OVEF

SUMMARY:
The main objective is to assess long term safety of treatment with oral nintedanib in patients with Systemic Sclerosis associated Interstitial Lung Disease (SSc-ILD).

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed the parent trial 1199.214/1199-0340 per protocol and did not permanently discontinue study treatment
* Signed and dated written informed consent in accordance with International Conference on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial
* Women of childbearing potential must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly as well as one barrier method for 28 days prior to nintedanib treatment initiation, during the trial and for 3 months after last intake of nintedanib.
* Further inclusion criteria apply

Exclusion Criteria:

* Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) > 3 x Upper Limit of Normal (ULN)
* Bilirubin > 2 x ULN
* Creatinine clearance <30 mL/min calculated by Cockcroft-Gault formula.
* Clinically relevant anaemia at investigators discretion.
* Bleeding risk, any of the following

  * Known genetic predisposition to bleeding according to the judgement of the investigator
  * Patients who require

    * Fibrinolysis, full-dose therapeutic anticoagulation
    * High dose antiplatelet therapy.
  * Hemorrhagic central nervous system (CNS) event after completion of the parent trial 1199.214/1199-0340
  * Any of the following after last treatment of 1199.214/1199-0340:

    * Haemoptysis or haematuria
    * Active gastro-intestinal bleeding or Gastrointestinal (GI) - ulcers
    * Gastric antral vascular ectasia (GAVE)
    * Major injury or surgery
  * Coagulation parameters: International normalised ratio (INR) >2, prolongation of prothrombin time (PT) and partial thromboplastin time (PTT) by >1.5 x ULN at Visit 1.
* New major thrombo-embolic events developed after completion of the parent trial 1199.214/1199-0340:

  * Stroke;
  * Deep vein thrombosis;
  * Pulmonary embolism;
  * Myocardial infarction.
* Major surgery performed within the next 3 months
* Time period > 12 weeks between last drug intake in 1199.214 or > 1 week between last nintedanib intake in trial 1199-0340 and Visit 2 of this trial
* Usage of any investigational drug after completion of 1199.214/1199-0340 or planned usage of an investigational drug during the course of this trial.
* A disease or condition which may put the patient at risk because of participation in this trial (e.g. clinically relevant intestinal pseudoobstruction) or limit the patient's ability to participate in this trial
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial subject or unlikely to complete the trial
* Known hypersensitivity to the trial medication or its components (i.e. soya lecithin).
* Women who are pregnant, nursing, or who plan to become pregnant while in the trial
* Previous enrolment in this trial
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (159):
- United States (39):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hospital for Special Surgery, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center-New York Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center - Vanderbilt Lung Institute at 100 Oaks, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Inova Fairfax Medical Campus, Falls Church, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Buenos Aires
  - APRILLUS-Asistencia e Investigación, Ciudad Autonoma Buenos Aires
  - CEMER-Centro Medico De Enfermedades Respiratorias, Florida
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Medical University of Innsbruck, Innsbruck, Austria
- Belgium (3):
  - UNIV UZ Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Edumed - Educacao e Saude SA, Curitiba, Brazil
- HSCM, Montreal, Quebec, Canada
- Chile (2):
  - Hospital Clínico Reg. de Concepción "Dr. G. Grant Benavente", Concepción
  - Centro de Investigación del Maule, Talca
- China (6):
  - Peking Union Medical College Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital, Chengdu
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huashan Hospital, Fudan University, Shanghai
  - The First Hospital of China Medical University, Shenyang
- Institute of Rheumathology Prague, Prague, Czechia
- Denmark (2):
  - Aarhus University Hospital, Aarhus N
  - Odense University Hospital, Odense
- Finland (2):
  - HYKS Keuhkosairauksien tutkimusyksikkö, Helsinki
  - TYKS, Turku
- France (12):
  - HOP Avicenne, Bobigny
  - HOP Louis Pradel, Bron
  - CHRU Lille, Lille
  - HOP Claude Huriez, Lille
  - HOP Arnaud de Villeneuve, Montpellier
  - HOP Hôtel-Dieu, Nantes
  - HOP Pasteur, Nice
  - HOP Bichat, Paris
  - HOP Pontchaillou, Rennes
  - HOP Charles Nicolle, Rouen
  - HOP Larrey, Toulouse
  - HOP Bretonneau, Tours
- Germany (10):
  - Klinik Donaustauf, Donaustauf
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Klinik Altona, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik-Heidelberg gGmbH am Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Münster, Münster
  - Universitätsklinikum Tübingen, Tübingen
- General Hospital of Athens "Laiko", Athens, Greece
- India (9):
  - Ramaiah Medical College and Hospitals, Bangalore
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Sir Gangaram Hospital, Delhi
  - Care Hospital, Hyderabad
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Asthma Bhawan, Jaipur
  - Getwell Hospital & Research Institute, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - B.J. Medical College and Sasoon General Hospital, Pune
- Israel (4):
  - Bnei Zion Medical Center, Haifa, Haifa
  - Rambam Medical Center, Haifa
  - Rabin Medical Center Beilinson, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Università degli Studi di Genova, Genova
  - A.O. San Gerardo di Monza, Monza
  - A.O Universitaria - Università degli Studi della Campania Luigi Vanvitelli, Napoli
  - Università degli Studi Padova, Padua
  - Azienda Universitaria-Universita' La Sapienza, Roma
- Japan (18):
  - Tosei General Hospital, Aichi, Seto
  - Kurume University Hospital, Fukuoka, Kurume
  - Sapporo Medical University Hospital, Hokkaido, Sapporo
  - National Hospital Organization Himeji Medical Center, Hyogo, Himeji
  - St. Marianna University Hospital, Kanagawa, Kawasaki
  - Kitasato University Hospital, Kanagawa, Sagamihara
  - Kanagawa Cardiovascular and Respiratory Center, Kanagawa, Yokohama
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Kindai University Hospital, Osaka, Osakasayama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Osaka, Sakai
  - Osaka Medical College Hospital, Osaka, Takatsuki
  - Saitama Medical University Hospital, Saitama, Iruma-gun
  - Hamamatsu University Hospital, Shizuoka, Hamamatsu
  - Tokushima University Hospital, Tokushima, Tokushima
  - Juntendo University Hospital, Tokyo, Bunkyo-Ku
  - Nippon Medical School Hospital, Tokyo, Bunkyo-Ku
  - Toho University Omori Medical Center, Tokyo, Ota-ku
  - Institute of Rheumatology Tokyo Women's Medical University, Tokyo, Shinjyuku-ku
- Malaysia (2):
  - Hospital Pulau Pinang, Georgetown Pulau Pinang
  - University of Malaya Medical Centre, Kuala Lumpur
- Instituto Nacional de Enfermedades Respiratorias Ismael Cosío Villegas, Mexico City, Mexico
- Netherlands (4):
  - Amsterdam UMC Locatie VUMC, Amsterdam
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Norway (2):
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (4):
  - Dr.Biziel UnivHosp#2,Rheumat&Connec.Tissue Disease,Bydgoszcz, Bydgoszcz
  - Specialist Allergy-Internist Center ALL-MED, Krakow
  - EMED, Center of Medical Services,Private Prac,Rzeszow, Rzeszów
  - Indep.Pblic Clin.Hosp#1,Dermatol,Venereol&Allerg.dep,Wroclaw, Wroclaw
- Portugal (6):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Fernando Fonseca, EPE, Amadora
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULSAM, EPE - Hospital Conde de Bertiandos, Ponte de Lima
  - Centro Hospitalar Universitário São João,EPE, Porto
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Spain (7):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Dr. Peset, Valencia
  - Hospital Politècnic La Fe, Valencia
  - Hospital Álvaro Cunqueiro, Vigo
- Clinical Rheumatology Research Center Sahlgrenska, Gothenburg, Sweden
- University Hospital Zurich, Zurich, Switzerland
- Thailand (3):
  - Ramathibodi Hospital, Bangkok
  - Srinagarind Hospital, Muang
  - Songklanagarind Hospital, Songkhla
- United Kingdom (4):
  - Royal Free Hospital, London
  - Guy's Hospital, London
  - Royal Brompton Hospital, London
  - Salford Royal Hospital, Salford

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Allanore Y, Khanna D, Smith V, Aringer M, Hoffmann-Vold AM, Kuwana M, Merkel PA, Stock C, Sambevski S, Denton CP; SENSCIS Trial Investigators. Effects of nintedanib in patients with limited cutaneous systemic sclerosis and interstitial lung disease. Rheumatology (Oxford). 2024 Mar 1;63(3):639-647. doi: 10.1093/rheumatology/kead280. PMID 37294870
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a prospective, open-label extension trial to assess long-term safety and tolerability of nintedanib in patients with Systemic Sclerosis associated Interstitial Lung Disease (SSc-ILD) who had completed treatment (including the follow-up visit or end of treatment/study visit, respectively) of the randomised, double-blind, placebo-controlled parent trial 1199.214 or trial 1199-0340.
Pre-assignment Details: Only patients with SSc-ILD who completed one of the parent trials on treatment (i.e., did not discontinue treatment early) were eligible and were included in this trial if they fulfilled all the inclusion criteria and did not present any of the exclusion criteria.
Period: Overall Study
Arm/Group | Nintedanib
Started | 444
Completed | 265
Not Completed | 179
Not completed — Adverse Event | 120
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 39
Not completed — Other than listed above | 15
Not completed — Covid-19 related | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): all patients who signed informed consent and received at least 1 dose of trial medication
Arm/Group | Nintedanib
Number analyzed (Participants) | 444
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335
  Male | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 406
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 110
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 18
  White | 308
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Any Adverse Event (AE) Over the Course of the Trial
Description: Number of patients with any adverse event (AE) over the course of the trial.
Time Frame: First trial medication intake up to last trial drug intake, plus 7 days residual effect period, up to approximate 60 months.
Population: Treated Set (TS): all patients who signed informed consent and received at least 1 dose of trial medication
Measure: Count of Participants; unit: Participants
Arm/Group | Nintedanib
Number analyzed (Participants) | 444
Participants | 441

ADVERSE EVENTS:
Time Frame: First trial medication intake up to last trial drug intake, plus 7 days residual effect period, up to ~59.9 months.
Description: Treated Set (TS): all patients who signed informed consent and received at least 1 dose of trial medication.
Arm/Group | Nintedanib
All-Cause Mortality (participants affected / at risk) | 23/444
Serious Adverse Events (participants affected / at risk) | 198/444
Other Adverse Events (participants affected / at risk) | 425/444
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=444)
Anaemia (Blood and lymphatic system disorders) | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Acute left ventricular failure (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 2
Atrial tachycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 7
Cardiac failure chronic (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Chordae tendinae rupture (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Left ventricular failure (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Pericarditis (Cardiac disorders) | 1
Right ventricular failure (Cardiac disorders) | 3
Sudden hearing loss (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Blindness unilateral (Eye disorders) | 1
Cataract (Eye disorders) | 2
Glaucoma (Eye disorders) | 2
Retinal detachment (Eye disorders) | 1
Retinal tear (Eye disorders) | 1
Vitreous detachment (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Pneumoperitoneum (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 1
Chest pain (General disorders) | 2
Disease progression (General disorders) | 1
General physical health deterioration (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 1
Polyserositis (General disorders) | 1
Pyrexia (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Drug-induced liver injury (Hepatobiliary disorders) | 4
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hydrocholecystis (Hepatobiliary disorders) | 1
Liver injury (Hepatobiliary disorders) | 5
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 2
Arthritis bacterial (Infections and infestations) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 9
COVID-19 pneumonia (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 1
Clostridium colitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 2
Diarrhoea infectious (Infections and infestations) | 2
Enteritis infectious (Infections and infestations) | 1
Escherichia infection (Infections and infestations) | 1
Gallbladder abscess (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Haemophilus infection (Infections and infestations) | 1
Infected bunion (Infections and infestations) | 1
Infected skin ulcer (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Intervertebral discitis (Infections and infestations) | 1
Labyrinthitis (Infections and infestations) | 1
Localised infection (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 3
Osteomyelitis (Infections and infestations) | 4
Pharyngotonsillitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 26
Pneumonia aspiration (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 3
Pneumonia mycoplasmal (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
Propionibacterium infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Subperiosteal abscess (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Animal bite (Injury, poisoning and procedural complications) | 1
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Spleen contusion (Injury, poisoning and procedural complications) | 1
Sternal fracture (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 1
Ejection fraction decreased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Hepatic enzyme increased (Investigations) | 1
Human metapneumovirus test positive (Investigations) | 1
Weight decreased (Investigations) | 3
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1
Crowned dens syndrome (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 4
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 1
Systemic scleroderma (Musculoskeletal and connective tissue disorders) | 2
Trismus (Musculoskeletal and connective tissue disorders) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Adenoid cystic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to gallbladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
T-cell type acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Cerebral haematoma (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Intracranial mass (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 13
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 7
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 17
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 1
Sclerema (Skin and subcutaneous tissue disorders) | 1
Scleroderma associated digital ulcer (Skin and subcutaneous tissue disorders) | 1
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 8
Arteriosclerosis (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Dry gangrene (Vascular disorders) | 2
Extremity necrosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral artery occlusion (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib (N=444)
Anaemia (Blood and lymphatic system disorders) | 24
Abdominal pain (Gastrointestinal disorders) | 52
Abdominal pain upper (Gastrointestinal disorders) | 24
Diarrhoea (Gastrointestinal disorders) | 338
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 43
Nausea (Gastrointestinal disorders) | 122
Vomiting (Gastrointestinal disorders) | 100
Fatigue (General disorders) | 46
Pyrexia (General disorders) | 28
Bronchitis (Infections and infestations) | 46
COVID-19 (Infections and infestations) | 68
Influenza (Infections and infestations) | 23
Nasopharyngitis (Infections and infestations) | 82
Respiratory tract infection (Infections and infestations) | 27
Upper respiratory tract infection (Infections and infestations) | 76
Urinary tract infection (Infections and infestations) | 43
Alanine aminotransferase increased (Investigations) | 47
Aspartate aminotransferase increased (Investigations) | 43
Gamma-glutamyltransferase increased (Investigations) | 33
Weight decreased (Investigations) | 63
Decreased appetite (Metabolism and nutrition disorders) | 33
Arthralgia (Musculoskeletal and connective tissue disorders) | 75
Back pain (Musculoskeletal and connective tissue disorders) | 41
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31
Dizziness (Nervous system disorders) | 24
Headache (Nervous system disorders) | 55
Cough (Respiratory, thoracic and mediastinal disorders) | 83
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47
Skin ulcer (Skin and subcutaneous tissue disorders) | 110
Hypertension (Vascular disorders) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT03313180/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT03313180/SAP_001.pdf